CLINICAL TRIAL: NCT05769777
Title: An Open-Label Multinational, Multicenter Study to Evaluate the Long-term Safety, Tolerability and Efficacy of Subcutaneous Amlitelimab in Participants Aged 12 Years and Older With Moderate to Severe Atopic Dermatitis
Brief Title: Open Label, Long-term Study Evaluating Safety and Efficacy of Subcutaneous Amlitelimab in Participants Aged 12 Years and Older With Moderate to Severe Atopic Dermatitis
Acronym: ATLANTIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS17789; U1111-1280-6080 (Other: ICTRP); 2022-502188-39 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Amlitelimab (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab

INTERVENTIONS:
Drug: Amlitelimab — Pharmaceutical form: Solution for injection; Route of administration: Subcutaneous (SC)

SUMMARY:
This is a single group, 1-arm, long-term safety study for treatment of participants with moderate to severe atopic dermatitis (AD).

The purpose of this study is to characterize the long-term safety and efficacy of amlitelimab in treated participants with age ≥12 years old with moderate to severe AD.

The study duration per participant will be up to 284 weeks, including:

* A screening period of up to 2 to 4 weeks
* An open label treatment period of up to 268 weeks (approximately 5 years)
* A post-treatment safety follow-up period of at least 20 weeks after the last dose administration (last IMP administration at Week 264)

The planned number of visits will be 35 visits.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 12 years of age inclusive, at the time of signing the informed consent.
* Participants must have AD as defined by the American Academy of Dermatology Consensus Criteria for 1 year or longer at baseline.
* Participant must have documented history (within 6 months prior to screening visit), of inadequate response (including inadequate efficacy or medical inadvisability) to topical treatments and/or inadequate response to systemic therapies (within 12 months prior to screening visit).
* Eczema Area Severity Index (EASI) of 16 or higher at baseline visit/Visit 2.
* Validated Investigator Global Assessment scale for atopic dermatitis (vIGA-AD) of 3 or 4 at baseline visit/Visit 2.
* AD involvement of 10% or more of body surface area (BSA) at baseline visit/Visit 2.
* Weekly average of daily Peak Pruritus-Numerical Rating Scale (PP-NRS) of ≥ 4 at baseline visit/Visit 2.
* Able and willing to comply with requested study visits and procedures.
* Body weight must be greater than or equal to 25 kg.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Female participants must not be pregnant or breastfeeding.

Exclusion Criteria:

* Skin co-morbidity that would adversely affect the ability to undertake AD assessments as per investigator's judgement
* Known history of or suspected significant current immunosuppression, including history of invasive opportunistic or helminthic infections despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged duration.
* Any malignancies or history of malignancies prior to baseline (except for non-melanoma skin cancer that has been excised and completely cured for more than 5 years prior to baseline).
* History of solid organ or stem cell transplant.
* Any pre-planned major elective surgery known about at baseline that in the opinion of the investigator would necessitate that IMP be permanently discontinued or require more than three doses to be missed.
* Severe concomitant illness that would in the Investigator's opinion inhibit the participant's participation in the study.
* Any medical or psychiatric condition which, in the opinion of the Investigator may present an unreasonable risk to the study participants as a result of his/her participation in this clinical study, may make participant's participation unreliable, or may interfere with study assessments.
* Any active or chronic infection including helminthic infection requiring systemic treatment within 4 weeks prior to baseline (1 week in the event of superficial skin infections); and any infection which as per Investigator's opinion precludes the participant's participation in the study.
* Treatment with live (attenuated) vaccines within 12 weeks prior to baseline; failure to complete non-live immunizations required by local regulation (eg, vaccination for COVID-19) at least 14 days prior to baseline.
* Having received any of the specified therapy within the specified timeframe(s) prior to the baseline visit.
* Positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C at the screening visit.
* Participants with active tuberculosis (TB), latent TB, a history of incompletely treated TB, suspected extrapulmonary TB infection, non-TB mycobacterial infection, or who are at high risk of contracting TB (such as close contact with individuals with active or latent TB) or received Bacillus Calmette-Guérin (BCG)-vaccination within 12 weeks prior to Screening.
* In the Investigator's opinion, any clinically significant laboratory results from the clinical chemistry, hematology, coagulation, or urinalysis tests at the screening visit.
* In the Investigator's opinion, any significant abnormality on 12-lead electrocardiogram (ECG) at the screening visit that could be suggestive of an unstable or underlying cardio-vascular condition that could preclude the participant's participation in the study.
* History of hypersensitivity or allergy to any of the excipients or IMP or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 901 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2031-06-11 (Estimated); Study Completion 2031-06-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who experienced Treatment-Emergent Adverse Events (TEAEs) | Baseline up to end of study (EOS) (Week 284)
  Percentage of participants who experienced TEAEs from baseline during the study
Percentage of participants who experienced Treatment-Emergent Serious Adverse Events (TESAEs) | Baseline up to EOS (Week 284)
  Percentage of participants who experienced TESAEs from baseline during the study

SECONDARY OUTCOMES:
Percentage of participants who experienced Treatment-Emergent Adverse Events of Special Interest (AESI) | Baseline up to EOS (Week 284)
  Percentage of participants who experienced AESI from baseline during the study
Percentage of participants with Potentially Clinically Significant Abnormalities (PCSA) for vital signs and clinical laboratory assessments, and electrocardiogram (ECG) | Baseline up to EOS (Week 284)
Percentage of participants discontinued from study treatment due to Adverse Events (AEs) | Baseline up to EOS (Week 284)
Percent change from baseline in Eczema Area and Severity Index (EASI) score | Baseline to EOS (Week 284)
  The EASI is an Investigator-assessed tool used to measure the extent (area) and severity of AD. The severity is assessed based on 4 disease characteristics (erythema, induration/papulation, excoriation and lichenification). The extent of involvement of AD is assessed in 4 body regions (head/neck, trunk, upper extremities and lower extremities). Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Proportion of participants with at least a 75% reduction from baseline in the EASI (EASI-75) | Baseline to EOS (Week 284)
Proportion of participants with at least a 50% reduction from baseline in the EASI (EASI-50) | Baseline to EOS (Week 284)
Proportion of participants with at least a 90% reduction from baseline in the EASI (EASI-90) | Baseline to EOS (Week 284)
Proportion of participants with at least 100% reduction from baseline in the EASI (EASI-100) | Baseline to EOS (Week 284)
Proportion of participants with Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD) of 0 (clear) or 1 (almost clear) and a reduction of ≥2 points from baseline | Baseline to EOS (Week 284)
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants with vIGA-AD 0 (clear) or 1 (almost clear) with presence of only barely perceptible erythema (no induration/papulation, no lichenification, no oozing or crusting) and a reduction from baseline of ≥2 points | Baseline to EOS (Week 284)
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Proportion of participants with vIGA-AD of 0 | Baseline to EOS (Week 284)
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Change in percent Body Surface Area (BSA) affected by AD from baseline | Baseline to EOS (Week 284)
  BSA affected by AD will measure the extent (area) of the disease.
Percent change in Scoring Atopic Dermatitis (SCORAD) index from baseline | Baseline to EOS (Week 284)
  The SCORAD Index is a clinical tool used to standardise the evaluation of the extent and severity of AD. To determine the extent of AD, the affected area (A) as a percentage of the whole body is determined, with a maximum score of 100%. The severity (B) of 6 specific symptoms of AD (redness, swelling, oozing/crusting, scratch marks, skin thickening [lichenification], dryness [area where there is no inflammation]) is assessed on a 4-point scale, with a maximum score of 18: none (0), mild (1), moderate (2) or severe (3). Subjective symptoms (C): itch and sleeplessness are recorded as scored by the participants or relative on a visual analogue scale (VAS), where 0 = no itch (or sleeplessness) and 10 = worst imaginable itch (or sleeplessness), with a maximum possible score of 20.
Proportion of participants requiring rescue treatment at each visit | Baseline to EOS (Week 284)
Proportion of participants with ≥4-point reduction in weekly average of daily Peak Pruritus-Numerical Rating Scale (PP-NRS) from baseline in participants with baseline weekly average of daily PP-NRS ≥4 | Baseline to EOS (Week 284)
  The PP-NRS is a single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD during the past 24 hours, with 0 = no itch and 10 = worst itch imaginable.
Proportion of participants with PP-NRS 0 or 1 | Baseline to EOS (Week 284)
  The PP-NRS is a single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD during the past 24 hours, with 0 = no itch and 10 = worst itch imaginable.
Percent change in weekly average of daily PP-NRS from baseline | Baseline to EOS (Week 284)
  The PP-NRS is a single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD during the past 24 hours, with 0 = no itch and 10 = worst itch imaginable.
Change in weekly average of daily Skin Pain-Numerical Rating Scale (SP-NRS) from baseline | Baseline to EOS (Week 284)
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD during the past 24 hours, with 0 = no pain and 10 = worst possible pain imaginable.
Proportion of participants with a reduction in weekly average of daily SP-NRS ≥4 from baseline in participants with baseline weekly average of daily SP-NRS ≥4 | Baseline to EOS (Week 284)
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD during the past 24 hours, with 0 = no pain and 10 = worst possible pain imaginable.
Change in weekly average of daily Sleep Disturbance-Numerical Rating Scale (SD-NRS) from baseline | Baseline to EOS (Week 284)
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD, with 0 being 'no sleep loss related to the symptoms of atopic dermatitis' and 10 being 'I did not sleep at all' due to the symptoms of atopic dermatitis".
Proportion of participants with a reduction in weekly average of daily SD-NRS ≥3 from baseline in participants with Baseline weekly average of daily SD-NRS ≥3 | Baseline to EOS (Week 284)
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD, with 0 being 'no sleep loss related to the symptoms of atopic dermatitis' and 10 being 'I did not sleep at all' due to the symptoms of atopic dermatitis".
Change in Patient Oriented Eczema Measure (POEM) from baseline | Baseline to EOS (Week 284)
  The POEM is a 7-item self-assessment questionnaire used for monitoring atopic eczema severity, focusing on the signs and symptoms as experienced by the patient during the past 7 days. Total score ranges from 0 to 28.
Proportion of participants with a reduction in POEM ≥4 from Baseline in participants with POEM baseline ≥4 | Baseline to EOS (Week 284)
  The POEM is a 7-item self-assessment questionnaire used for monitoring atopic eczema severity, focusing on the signs and symptoms as experienced by the patient during the past 7 days. Total score ranges from 0 to 28.
Proportion of adolescent participants with a reduction in POEM ≥6 from Baseline in adolescents with POEM baseline ≥6 | Baseline to EOS (Week 284)
  The POEM is a 7-item self-assessment questionnaire used for monitoring atopic eczema severity, focusing on the signs and symptoms as experienced by the patient during the past 7 days. Total score ranges from 0 to 28.
Change in Atopic Dermatitis Control Test (ADCT) from baseline | Baseline to EOS (Week 284)
  The ADCT is a 6-item patient-reported outcomes instrument with a 7-day recall period to measure AD disease control. Total score ranges from 0 to 24.
Proportion of participants with a reduction in ADCT ≥5 from baseline in participants with baseline ADCT≥7 | Baseline to EOS (Week 284)
  The ADCT is a 6-item patient-reported outcomes instrument with a 7-day recall period to measure AD disease control. Total score ranges from 0 to 24.
Change in Dermatology Quality of Life Index (DLQI) from baseline in participants with age ≥16 years old | Baseline to EOS (Week 284)
  The DLQI is a 10-item questionnaire to measure dermatology specific quality of life (QoL), covering the participant's previous week (i.e. past 7 days). Total score ranges from 0 to 30, with higher scores indicating greater detrimental impact on QoL.
Change in Children's Dermatology Life Quality Index (CDLQI) from baseline in participants with age ≥12 to <16 years old | Baseline to EOS (Week 284)
  The CDLQI is a 10-item questionnaire to assess the impact of skin disease on a child's health related quality of life (HRQoL) over a recall period of 1 week. It is validated in children aged 4 to <16 years. Total score ranges from 0 to 30, with higher scores indicating greater detrimental impact on QoL.
Proportion of participants with age ≥12 to <16 with a reduction in CDLQI ≥4 from Baseline in participants with age ≥12 to <16 years old with CDLQI at baseline ≥6 | Baseline to EOS (Week 284)
  The CDLQI is a 10-item questionnaire to assess the impact of skin disease on a child's health related quality of life (HRQoL) over a recall period of 1 week. It is validated in children aged 4 to <16 years. Total score ranges from 0 to 30, with higher scores indicating greater detrimental impact on QoL.
Proportion of participants with age ≥12 to <16 with a reduction in CDLQI ≥6 from Baseline in participants with age ≥12 to <16 years old with CDLQI at baseline ≥6 | Baseline to EOS (Week 284)
  The CDLQI is a 10-item questionnaire to assess the impact of skin disease on a child's health related quality of life (HRQoL) over a recall period of 1 week. It is validated in children aged 4 to <16 years. Total score ranges from 0 to 30, with higher scores indicating greater detrimental impact on QoL.
Proportion of participants with a reduction in DLQI ≥4 from Baseline in participants with age ≥16 years old and with DLQI at baseline ≥4 | Baseline to EOS (Week 284)
  The DLQI is a 10-item questionnaire to measure dermatology specific quality of life (QoL), covering the participant's previous week (i.e. past 7 days). Total score ranges from 0 to 30, with higher scores indicating greater detrimental impact on QoL.
Change in Patient Global Impression of Severity (PGIS) from baseline | Baseline to EOS (Week 284)
  The PGIS is a single item tool used to assess current severity of eczema symptoms, scored on a 5-point scale from 1 = no symptoms to 5 = very severe symptoms.
Proportions of participants who report symptoms to be "No" on the PGIS score | Baseline to EOS (Week 284)
  The PGIS is a single item tool used to assess current severity of eczema symptoms, scored on a 5-point scale from 1 = no symptoms to 5 = very severe symptoms.
Proportions of participants who report symptoms to be "No" or "Mild" on the PGIS score | Baseline to EOS (Week 284)
  The PGIS is a single item tool used to assess current severity of eczema symptoms, scored on a 5-point scale from 1 = no symptoms to 5 = very severe symptoms.
Proportion of participants who respond "Much better" on the Patient Global Impression of (PGIC) scale | Week 16 to EOS (Week 284)
  The PGIC is a single item global tool used in the assessment of AD, scored on a 5-point scale from 1 = Much improved to 5 = Much worse.
Proportion of participants who respond "Much better" or "A little better" on the PGIC scale | Week 16 to EOS (Week 284)
  The PGIC is a single item global tool used in the assessment of AD, scored on a 5-point scale from 1 = Much improved to 5 = Much worse.
Proportion of participants by PGIC responses | Week 16 to EOS (Week 284)
  The PGIC is a single item global tool used in the assessment of AD, scored on a 5-point scale from 1 = Much improved to 5 = Much worse.
Change in Hospital Anxiety Depression Scale (HADS) from baseline | Baseline to EOS (Week 284)
  The HADS is a 14-item patient-reported outcomes measure used to assess states of anxiety and depression over the past week. It is comprised of 7 items assessing anxiety and depression respectively. A Total score is out of 42 (21 per subscale). Higher scores indicate greater levels of anxiety and/or depression.
Proportion of participants with HADS subscale Anxiety (HADS-A) <8 in participants with baseline HADS-A ≥8 | Baseline to EOS (Week 284)
  The HADS is a 14-item patient-reported outcomes measure used to assess states of anxiety and depression over the past week. It is comprised of 7 items assessing anxiety and depression respectively. A Total score is out of 42 (21 per subscale). Higher scores indicate greater levels of anxiety and/or depression.
  HADS-A is the anxiety HADS subscale.
Proportion of participants with HADS subscale Depression (HADS-D) <8 in participants with HADS-D Baseline ≥8 | Baseline to EOS (Week 284)
  The HADS is a 14-item patient-reported outcomes measure used to assess states of anxiety and depression over the past week. It is comprised of 7 items assessing anxiety and depression respectively. A Total score is out of 42 (21 per subscale). Higher scores indicate greater levels of anxiety and/or depression.
  HADS-D is the depression HADS subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (176):
- United States (23):
  - Allervie Clinical Research - Birmingham- Site Number : 8400050, Birmingham, Alabama
  - Research Solutions of Arizona- Site Number : 8400020, Litchfield Park, Arizona
  - Dermatology Trial Associates- Site Number : 8400027, Bryant, Arkansas
  - University Dermatology Trials- Site Number : 8400052, Newport Beach, California
  - Children's Hospital Colorado - Aurora- Site Number : 8400041, Aurora, Colorado
  - IMMUNOe International Research Centers - Centennial- Site Number : 8400024, Centennial, Colorado
  - Renaissance Research and Medical Group- Site Number : 8400006, Cape Coral, Florida
  - Florida Pharmaceutical Research and Associates- Site Number : 8400018, Miami, Florida
  - Miami Clinical Research Tower- Site Number : 8400036, Miami, Florida
  - Florida Research Center- Site Number : 8400011, Miami, Florida
  - Bio-Medical Research- Site Number : 8400037, Miami, Florida
  - Clinical Research Trials of Florida- Site Number : 8400054, Tampa, Florida
  - Advanced Medical Research - Atlanta- Site Number : 8400044, Atlanta, Georgia
  - Georgia Skin & Cancer Clinic- Site Number : 8400048, Savannah, Georgia
  - Sneeze Wheeze & Itch Associates- Site Number : 8400002, Normal, Illinois
  - Kentucky Advanced Medical Research- Site Number : 8400014, Murray, Kentucky
  - The Derm Institute of West Michigan- Site Number : 8400043, Caledonia, Michigan
  - Michigan Dermatology Institute - Livonia- Site Number : 8401010, Livonia, Michigan
  - Michigan Dermatology Institute - Waterford- Site Number : 8400010, Waterford, Michigan
  - Dermatology Research Center of Oklahoma- Site Number : 8400035, Tulsa, Oklahoma
  - The Children's Hospital of Philadelphia- Site Number : 8400009, Philadelphia, Pennsylvania
  - Texas Dermatology and Laser Specialists - San Antonio - Oakwell Court- Site Number : 8400053, San Antonio, Texas
  - Private Practice - Dr. Marthe N. Dika- Site Number : 8400022, Burlington, Wisconsin
- Argentina (10):
  - Investigational Site Number : 0320022, General Pico, La Pampa Province
  - Investigational Site Number : 0320006, Rosario, Santa Fe Province
  - Investigational Site Number : 0320007, Rosario, Santa Fe Province
  - Investigational Site Number : 0320008, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320003, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320009, Buenos Aires
  - Investigational Site Number : 0320005, Buenos Aires
- Australia (2):
  - Investigational Site Number : 0360002, Kogarah, New South Wales
  - Investigational Site Number : 0360001, Sydney, New South Wales
- Brazil (9):
  - Centro de Pesquisas da Clínica IBIS- Site Number : 0760002, Salvador, Estado de Bahia
  - Hospital de Clinicas da Universidade Federal do Parana- Site Number : 0760022, Curitiba, Paraná
  - Pontifica Universidade Catolica do Parana- Site Number : 0760023, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre- Site Number : 0760005, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto- Site Number : 0760008, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC- Site Number : 0760001, Santo André, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto- Site Number : 0760003, São José do Rio Preto, São Paulo
  - Clinica de Alergia Martti Antila- Site Number : 0760006, Sorocaba, São Paulo
  - IDERJ - Instituto de Dermatologia e Estética do Brasil- Site Number : 0760004, Rio de Janeiro
- Canada (13):
  - Investigational Site Number : 1240001, Calgary, Alberta
  - Investigational Site Number : 1240052, Edmonton, Alberta
  - Investigational Site Number : 1240051, Vancouver, British Columbia
  - Investigational Site Number : 1240009, Etobicoke, Ontario
  - Investigational Site Number : 1240008, Mississauga, Ontario
  - Investigational Site Number : 1240011, Oakville, Ontario
  - Investigational Site Number : 1240004, Peterborough, Ontario
  - Investigational Site Number : 1240003, Richmond Hill, Ontario
  - Investigational Site Number : 1240012, Toronto, Ontario
  - Investigational Site Number : 1240002, Montreal, Quebec
  - Investigational Site Number : 1240010, Québec, Quebec
  - Investigational Site Number : 1240006, Québec, Quebec
  - Investigational Site Number : 1240044, Saskatoon, Saskatchewan
- Chile (11):
  - Investigational Site Number : 1520004, Valdivia, Los Ríos Region
  - Investigational Site Number : 1520013, Lo Barnechea, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520009, Osorno, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520011, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520008, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520010, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520014, Chillán
- China (16):
  - Investigational Site Number : 1560015, Beijing
  - Investigational Site Number : 1560008, Changchun
  - Investigational Site Number : 1560016, Changsha
  - Investigational Site Number : 1560014, Chengdu
  - Investigational Site Number : 1560072, Fuzhou
  - Investigational Site Number : 1560074, Guangzhou
  - Investigational Site Number : 1560044, Hangzhou
  - Investigational Site Number : 1560013, Jingzhou
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560018, Suzhou
  - Investigational Site Number : 1560010, Taiyuan
  - Investigational Site Number : 1560073, Taizhou
  - Investigational Site Number : 1560019, Xinxiang
  - Investigational Site Number : 1560012, Yinchuan
  - Investigational Site Number : 1560011, Yiwu
  - Investigational Site Number : 1560028, Zhenjiang
- Czechia (6):
  - Investigational Site Number : 2032105, Nový Jičín
  - Investigational Site Number : 2032104, Ostrava
  - Investigational Site Number : 2032102, Prague
  - Investigational Site Number : 2030003, Prague
  - Investigational Site Number : 2030006, Prague
  - Investigational Site Number : 2030007, Prague
- Investigational Site Number : 2080001, Aarhus, Denmark
- France (7):
  - Investigational Site Number : 2500004, Créteil
  - Investigational Site Number : 2500001, Lille
  - Investigational Site Number : 2500005, Marseille
  - Investigational Site Number : 2500009, Nantes
  - Investigational Site Number : 2500003, Paris
  - Investigational Site Number : 2500006, Pierre-Bénite
  - Investigational Site Number : 2500002, Toulouse
- Germany (5):
  - Investigational Site Number : 2760009, Bad Bentheim
  - Investigational Site Number : 2762203, Berlin
  - Investigational Site Number : 2762205, Dresden
  - Investigational Site Number : 2762201, Münster
  - Investigational Site Number : 2760010, Osnabrück
- India (7):
  - Investigational Site Number : 3560006, Bengaluru
  - Investigational Site Number : 3560007, Bikaner
  - Investigational Site Number : 3560011, Kochi
  - Investigational Site Number : 3560005, Kolkata
  - Investigational Site Number : 3560004, Mangaluru
  - Investigational Site Number : 3560002, Nashik
  - Investigational Site Number : 3560008, Surat
- Italy (7):
  - Investigational Site Number : 3800003, Milan, Milano
  - Investigational Site Number : 3800002, Naples, Napoli
  - Investigational Site Number : 3800004, Naples, Napoli
  - Investigational Site Number : 3800007, Rome, Roma
  - Investigational Site Number : 3800006, Rome, Roma
  - Investigational Site Number : 3800005, Brescia
  - Investigational Site Number : 3800008, Vicenza
- Japan (5):
  - Investigational Site Number : 3923114, Obihiro, Hokkaido
  - Investigational Site Number : 3923113, Yokohama, Kanagawa
  - Investigational Site Number : 3923110, Sakai, Osaka
  - Investigational Site Number : 3923106, Mibu, Tochigi
  - Investigational Site Number : 3920001, Tachikawa, Tokyo
- Mexico (2):
  - Investigational Site Number : 4840001, Chihuahua City
  - Investigational Site Number : 4840008, Durango
- Netherlands (3):
  - Investigational Site Number : 5280002, Breda
  - Investigational Site Number : 5280004, Rotterdam
  - Investigational Site Number : 5280001, Utrecht
- Poland (8):
  - Investigational Site Number : 6160014, Lodz, Lódzkie
  - Investigational Site Number : 6162411, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160009, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160007, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160006, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number : 6160001, Chorzów, Silesian Voivodeship
  - Investigational Site Number : 6160003, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160012, Lublin
- Caribbean Medical Research Center- Site Number : 8400028, San Juan, Puerto Rico
- South Africa (12):
  - Investigational Site Number : 7100011, Cape Town
  - Investigational Site Number : 7100010, Cape Town
  - Investigational Site Number : 7100002, Cape Town
  - Investigational Site Number : 7100009, Cape Town
  - Investigational Site Number : 7100012, Durban
  - Investigational Site Number : 7100015, Durban
  - Investigational Site Number : 7100007, Johannesburg
  - Investigational Site Number : 7100006, Kempton Park
  - Investigational Site Number : 7100005, Middelburg
  - Investigational Site Number : 7100003, Pretoria
  - Investigational Site Number : 7100014, Pretoria
  - Investigational Site Number : 7100004, Reiger Park
- South Korea (6):
  - Investigational Site Number : 4100002, Ansan-si, Gyeonggi-do
  - Investigational Site Number : 4100016, Bucheon-si, Gyeonggi-do
  - Investigational Site Number : 4100003, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 4100018, Incheon, Incheon-gwangyeoksi
  - Investigational Site Number : 4100006, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
- Spain (6):
  - Investigational Site Number : 7240002, Badalona, Barcelona [Barcelona]
  - Investigational Site Number : 7240022, Sabadell, Barcelona [Barcelona]
  - Investigational Site Number : 7242505, Alicante
  - Investigational Site Number : 7242501, Córdoba
  - Investigational Site Number : 7242503, Madrid
  - Investigational Site Number : 7240006, Valencia
- Investigational Site Number : 7560002, Buochs, Switzerland
- Taiwan (7):
  - Investigational Site Number : 1580006, Hsinchu
  - Investigational Site Number : 1583201, Kaohsiung City
  - Investigational Site Number : 1580002, New Taipei City
  - Investigational Site Number : 1583202, Taichung
  - Investigational Site Number : 1580007, Taichung
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1583203, Taoyuan
- Turkey (Türkiye) (4):
  - Investigational Site Number : 7920002, Aydin
  - Investigational Site Number : 7920003, İzmit
  - Investigational Site Number : 7920005, Manisa
  - Investigational Site Number : 7920004, Trabzon
- United Kingdom (4):
  - Investigational Site Number : 8260001, London, England
  - Investigational Site Number : 8262601, London, London, City of
  - Investigational Site Number : 8260002, Edinburgh
  - Investigational Site Number : 8260004, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LTS17789 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25307&tenant=MT_SNY_9011